CLINICAL TRIAL: NCT04514107
Title: A Cluster-Randomized Trial to Evaluate the Efficacy of Wolbachia-Infected Aedes Aegypti Mosquitoes in Reducing the Incidence of Arboviral Infection in Brazil
Brief Title: A Cluster-randomized Trial to EValuate the Efficacy of Wolbachia-InfecTed Aedes Aegypti Mosquitoes in Reducing the Incidence of Arboviral Infection in Brazil (EVITA Dengue)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-0111; HHSN272201300018I
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-05-29

CONDITIONS: Dengue Fever
Keywords: Arbovirus; Brazil; Chikungunya; Cluster-Randomized; Dengue; Flavivirus; Mosquitoes; Wolbachia-infected; Zika virus
MeSH Terms: conditions — Dengue; Chikungunya Fever; Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): 29 school-based clusters of healthy individuals, age 6-11, exposed to standard vector control efforts recommended by the Brazilian National Dengue Control Program (PNCD). n=1740
  Interventions: Other: Brazilian National Dengue Control Program
- Intervention (Experimental): 29 school-based clusters of healthy individuals, age 6-11, exposed to standard vector control efforts recommended by the Brazilian National Dengue Control Program (PNCD) and Wolbachia-infected Aedes aegypti (wMel) mosquitoes. n=1740
  Interventions: Other: Brazilian National Dengue Control Program; Other: Wolbachia-infected Aedes aegypti

INTERVENTIONS:
Other: Brazilian National Dengue Control Program — This program has 4 basic principles: 1) Adequate case finding, classification and treatment; 2) Epidemiological surveillance and reporting of all cases; 3) Mobilization and communication of risks to the public; 4) mosquito monitoring and control which consists fundamentally of detection of larva using a rapid larval index (LIRAa) followed by removal of breeding sites and local spraying.
Other: Wolbachia-infected Aedes aegypti — Brazilian strain of Aedes aegypti infected with Wolbachia pipientis released into geographic clusters.
  Arms: Intervention

SUMMARY:
This is a cluster randomized controlled trial (CRCT) to evaluate the efficacy of Wolbachia-infected A. aegypti mosquito releases in reducing the burden of ARBV infection in Brazil over four years. The intervention will be the release of Wolbachia-infected A. aegypti mosquitoes. Standard control measures routinely established by the Belo Horizonte City Hall as recommended by the PNCD, will continue to be performed by the Belo Horizonte Health Department (Zoonoses Management) in all clusters, that is, the standard control measures will be carried out throughout the city of Belo Horizonte, independent of this clinical study. Wolbachia-infected A. aegypti will be deployed by releasing adult mosquitoes in pre-determined, thoroughly spaced release points in easily accessible roads described in a release map. A release map will be generated for each cluster and the numbers of release points will be determined by population density, surface area and mosquito abundance. Wolbachia-infected A. aegypti mosquitoes will be deployed across intervention clusters in two stages: 1) a 4 month establishment stage in which most of the releases will occur and 2) followed by an 8 month consolidation stage in which the abundance of Wolbachia-infected mosquitoes will be measured and remedial deployments will be completed, if needed, with the aim of achieving a high prevalence of Wolbachia amongst A. aegypti mosquitoes in intervention clusters within 12 months from the start of the release. The goal is to reach a Wolbachia prevalence of 60% or higher. Monitoring of Wolbachia prevalence in the cluster will continue throughout the study period, but no further mosquito deployments will occur after the consolidation stage is complete. The primary objective is to evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of ARBV infection compared to standard Aedes vector control measures alone.

DETAILED DESCRIPTION:
This is a cluster randomized controlled trial (CRCT) to evaluate the efficacy of Wolbachia-infected A. aegypti mosquito releases in reducing the burden of ARBV infection in Brazil over four years. The intervention will be the release of Wolbachia-infected A. aegypti mosquitoes. Standard control measures routinely established by the Belo Horizonte City Hall as recommended by the PNCD, will continue to be performed by the Belo Horizonte Health Department (Zoonoses Management) in all clusters, that is, the standard control measures will be carried out throughout the city of Belo Horizonte, independent of this clinical study. Wolbachia-infected A. aegypti will be deployed by releasing adult mosquitoes in pre-determined, thoroughly spaced release points in easily accessible roads described in a release map. A release map will be generated for each cluster and the numbers of release points will be determined by population density, surface area and mosquito abundance. Wolbachia-infected A. aegypti mosquitoes will be deployed across intervention clusters in two stages: 1) a 4 month establishment stage in which most of the releases will occur and 2) followed by an 8 month consolidation stage in which the abundance of Wolbachia-infected mosquitoes will be measured and remedial deployments will be completed, if needed, with the aim of achieving a high prevalence of Wolbachia amongst A. aegypti mosquitoes in intervention clusters within 12 months from the start of the release. The goal is to reach a Wolbachia prevalence of 60% or higher. Monitoring of Wolbachia prevalence in the cluster will continue throughout the study period, but no further mosquito deployments will occur after the consolidation stage is complete.

Of note, due to widespread dengue epidemic in Brazil and the introduction of the dengue vaccination campaign by the Ministry of Health, all children ages 10-14 received Odenga. Since vaccination precludes the ability to assess for flavivirus seroconversion, participants eligible to receive the vaccination, the Year 5 annual sample may be collected earlier than the study window. The Visit 05 sample for these subjects will be obtained prior or up to 14 days after dengue vaccination (the optimal cut-off time for the detection of vaccine-induced neutralizing antibodies is to be determined and will be explained in more detail in the SAP). Those who have this earlier visit will also have Visit 06 during the expected study window. The Visit 06 sample will be used for serologic assay wherever available and appropriate considering dengue vaccination status and Visit 05 samples in all other circumstances.

The primary objective is to evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduce the sero-incidence of ARBV infection compared to standard Aedes vector control measures alone. The Secondary objectives are 1.) To evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of ARBV infection, inferred from model-based reconstruction of serological dynamics compared to standard Aedes vector control measures alone; 2.) To evaluate whether releases of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of FLAV or CHIKV infection amongst individuals who are seronegative to each of these viruses, respectively, at study entry, compared to standard Aedes vector control measures alone; 3.) To evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the overall sero-incidence of FLAV (DENV + ZIKV) infection; 4.) To evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of DENV infection; 5.) To evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of ZIKV infection; 6.) To evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of CHIKV infection among those who are CHIKV seronegative at baseline; 7.) To evaluate whether release of Wolbachia-infected Aedes aegypti mosquitoes plus standard Aedes vector control measures reduces the sero-incidence of DENV infection amongst individuals who are seropositive to any DENV serotype(s) at study entry, compared to standard Aedes vector control measures alone; 8.) To use model-based geostatistics to estimate the proportion and abundance of Wolbachia-infected and wildtype Aedes aegypti mosquitoes in intervention clusters during the study period; 9.) To use model-based geostatistics to estimate the proportion and abundance of Wolbachia-infected and wildtype Aedes aegypti mosquitoes in control clusters during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-11 years at enrollment.
2. Child's parent or legal guardian agrees to provide written informed consent.
3. Child agrees to provide informed assent.
4. Child is enrolled in a public school selected for this trial (and which define the clusters).
5. Child resides within geographic boundaries at least 5 days a week in the cluster area corresponding to his/her school.

Exclusion Criteria:

1. Children planning to move outside of the cluster boundary within the study period.
2. Child has poor venous access.
3. Child has received an experimental or licensed vaccine against dengue, Zika or chikungunya at enrollment. Participants who received a dengue, Zika or CHIK vaccine after enrollment will not be excluded.
4. Child has any medical condition that would prevent them from completing a blood draw.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5757 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Incidence of arbovirus (ARBV) infection | Year 1 through Year 5
  Defined as seroconversion to flavivirus (FLAV) or chikungunya virus (CHIKV), as detected during annual serological evaluations.

SECONDARY OUTCOMES:
Cluster level of prevalence and abundance of Wolbachia-infected and wildtype Aedes aegypti adults in control clusters | From Year 1 through Year 5
  As estimated by analysis of trap level data
Cluster level prevalence and abundance of Wolbachia-infected and wildtype Aedes aegypti adults in intervention clusters | From Year 1 through Year 5
  As estimated by analysis of trap level data
Incidence of arbovirus (ARBV) infections, specifically due to flavivirus (FLAV) or chikungunya virus (CHIKV) | Year 1 through Year 5
  As detected during annual serological evaluations; inferred from model-based reconstruction of serological dynamics
Incidence of Chikungunya virus (CHIKV) infection is defined by seroconversion to CHIKV | Year 1 through Year 5
  As detected during annual serological evaluations
Incidence of Dengue virus (DENV) infection as defined by seroconversion to DENV | Year 1 through Year 5
  As detected during annual serological evaluations
Incidence of Dengue virus (DENV) infection is defined by seroconversion | Year 1 through Year 5
  As detected during annual serological evaluations in the subgroup of participants who are seropositive at baseline (time of enrollment) to any DENV serotype(s) regardless of Zika Virus (ZIKV) serostatus
Incidence of Flavivirus (FLAV) infection as defined by seroconversion to FLAV | Year 1 through Year 5
  As detected during annual serological evaluations
Incidence of Zika virus (ZIKV) infection is defined as seroconversion to ZIKV | Year 1 through Year 5
  As detected during annual serological evaluations
Incident Arbovirus (ARBV) infections, as defined by seroconversion to Flavivirus (FLAV) | Year 1 through Year 5
  Among the subgroup of participants who have a Focus Reduction Neutralization Test (FRNT) 50 titer <1:20 at the baseline survey (time of enrollment) OR seroconversion to chikungunya virus (CHIKV)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Minas Gerais, Instituto de Ciencias Biologicas, Department of Biochemistry and Immunology, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Collins MH, Potter GE, Hitchings MDT, Butler E, Wiles M, Kennedy JK, Pinto SB, Teixeira ABM, Casanovas-Massana A, Rouphael NG, Deye GA, Simmons CP, Moreira LA, Nogueira ML, Cummings DAT, Ko AI, Teixeira MM, Edupuganti S. EVITA Dengue: a cluster-randomized controlled trial to EValuate the efficacy of Wolbachia-InfecTed Aedes aegypti mosquitoes in reducing the incidence of Arboviral infection in Brazil. Trials. 2022 Mar 2;23(1):185. doi: 10.1186/s13063-022-05997-4. PMID 35236394

DOCUMENTS (1):
  • Informed Consent Form (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04514107/ICF_000.pdf